CLINICAL TRIAL: NCT04981938
Title: Perfusion and Functional Results After Pulmonary Artery Reconstruction During Oncologic Lung Resection
Brief Title: Pulmonary Function After Arterial Sleeve Lobectomy
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Universitaire Montpellier (Other)
Responsible Party: Principal Investigator, Aude NGUYEN, Thoracic surgery resident, Centre Hospitalier Régional Universitaire Montpellier
Other Study IDs: CHRUMontpellier
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-07

CONDITIONS: Lung Cancer, Nonsmall Cell
Keywords: artery pulmonary reconstruction; sleeve lobectomy; lobectomy with angioplasty; arterial sleeve lobectomy; pulmonary function
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lobectomy with angioplasty: 81 patients who underwent lobectomy with pulmonary artery reconstruction during oncologic lung resection from January 2001 to December 2020
  Interventions: Procedure: Lobectomy with pulmonary artery reconstruction

INTERVENTIONS:
Procedure: Lobectomy with pulmonary artery reconstruction — Lobectomy with pulmonary artery reconstruction under general anesthesia with selective intubation, by postero-lateral thoracotomy in the fifth intercostal space
  Subgroups : different types of pulmonary artery reconstruction such as :
  * Tangential vascular reconstruction with direct suture
  * Circumferential resection and end-to-end anastomosis
  * bypass reconstruction with heterologous biografts, synthetic grafts, or pericardium patch

SUMMARY:
Lung cancer is the leading cause of cancer death worldwide. Despite the evolution of medical and multimodal treatments, surgical treatment remains the curative management in the localized cancer.

Historically, in central lung tumors, pneumonectomy was the gold standard. Currently, bronchial sleeve lobectomy is recommended as first-line treatment over pneumonectomy when complete resection is possible (Grade 2C).

In the case of pulmonary artery invasion, lobectomy with arterial resection and reconstruction is now an accepted option for central localized cancer.

Despite surgical challenge, arterial sleeve lobectomy is oncologically comparable with pneumonectomy while avoiding the high morbi-mortality.

Indeed, this surgery has shown better results than pneumonectomy in terms of overall survival, post-operative mortality, and quality of life.

Initially performed in patients with impaired cardio-pulmonary reserves, this parenchymal sparing procedure can be realised in all patients, when anatomical conditions allow a complete resection.

In the literature, no study has yet specifically investigated postoperative respiratory function after arterial sleeve lobectomy.

The investigators designed a retrospective monocentric study at the University Hospital of Montpellier on 81 lobectomies with pulmonary artery sleeve resection for lung cancer, from January 2001 to December 2020.

ELIGIBILITY:
Inclusion Criteria:

* all major lung resection with pulmonary artery reconstruction for lung cancer
* from January 2001 to December 2020 at University Hospital of Montpellier
* patient > 18 years

Exclusion Criteria:

0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes 81 patients: 18 womens, 63 mens There was no significant difference in patient characteristics.
  The most common resection was left upper lobectomy (52/81). 61 patients had a lung cancer with invasion of the left pulmonary artery.
  The most common histology was squamous cell carcinoma (42/81). 28 patients underwent a double sleeve (angioplasty and bronchoplasty)
  The type of arterial reconstruction was distributed as follows:
  * 25 bypass
  * 17 patch angioplasty
  * 16 circumferential resection and end-to-end anastomosis
  * 23 tangential vascular reconstruction with direct suture
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Impact of pulmonary artery reconstruction on perfusion on the remaining lung lobe (ventilation/perfusion scan) | 2001-2020
  Comparison of perfusion data on pre and post operative ventilation/perfusion scan

SECONDARY OUTCOMES:
Impact of pulmonary artery reconstruction on pulmonary function | 2001-2020
  Comparison of post operative predicted FEV1 to post operative FEV1
pulmonary artery reconstruction patency | 2001-2020
  Patency data of the arterial reconstruction (thoracic angioscan)
Pulmonary function according to the type of reconstruction | 2001-2020
  Comparison of the results (FEV1 ans patency) according to the type of reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: SOLOVEI Laurence, Principal Investigator — University Hospital, Montpellier
Locations (1):
- NGUYEN, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] D'Andrilli A, Maurizi G, Andreetti C, Ciccone AM, Ibrahim M, Poggi C, Venuta F, Rendina EA. Pulmonary artery reconstruction with pulmonary vein conduit for lung cancer: medium-term results. Ann Thorac Surg. 2014 Sep;98(3):990-5. doi: 10.1016/j.athoracsur.2014.04.110. Epub 2014 Jul 16. PMID 25038016
- [Background] D'Andrilli A, Maurizi G, Ciccone AM, Andreetti C, Ibrahim M, Menna C, Vanni C, Venuta F, Rendina EA. Long-segment pulmonary artery resection to avoid pneumonectomy: long-term results after prosthetic replacement. Eur J Cardiothorac Surg. 2018 Feb 1;53(2):331-335. doi: 10.1093/ejcts/ezx353. PMID 29029026
- [Background] Cerezo F, Cano JR, Espinosa D, Salvatierra A. New technique for pulmonary artery reconstruction. Eur J Cardiothorac Surg. 2009 Aug;36(2):422-3. doi: 10.1016/j.ejcts.2009.03.060. Epub 2009 Jun 5. PMID 19501519
- [Background] Cerfolio RJ, Bryant AS. Surgical techniques and results for partial or circumferential sleeve resection of the pulmonary artery for patients with non-small cell lung cancer. Ann Thorac Surg. 2007 Jun;83(6):1971-6; discussion 1976-7. doi: 10.1016/j.athoracsur.2007.01.048. PMID 17532380
- [Background] Galetta D, Borri A, Gasparri R, Petrella F, Spaggiari L. Surgical Techniques and Long-Term Results of Pulmonary Artery Reconstruction in Patients With Lung Cancer. Ann Thorac Surg. 2015 Oct;100(4):1196-202; discussion 1202. doi: 10.1016/j.athoracsur.2015.04.124. Epub 2015 Jul 21. PMID 26209482
- [Background] Gomez-Caro A, Martinez E, Rodriguez A, Sanchez D, Martorell J, Gimferrer JM, Haverich A, Harringer W, Pomar JL, Macchiarini P. Cryopreserved arterial allograft reconstruction after excision of thoracic malignancies. Ann Thorac Surg. 2008 Dec;86(6):1753-61; discussion 1761. doi: 10.1016/j.athoracsur.2008.06.027. PMID 19021970
- [Background] Ma Q, Liu D, Guo Y, Shi B, Tian Y, Song Z, Zhang Z, Ge B, Wang X, D'Amico TA. Surgical techniques and results of the pulmonary artery reconstruction for patients with central non-small cell lung cancer. J Cardiothorac Surg. 2013 Dec 1;8:219. doi: 10.1186/1749-8090-8-219. PMID 24289720
- [Background] Madariaga MLL, Geller A, Lanuti M, Ott H, Allan JS, Donahue DM, Mathisen DJ, Wright CD, Gaissert HA. Pulmonary Artery Resection During Lung Resection for Malignancy. Ann Thorac Surg. 2019 Dec;108(6):1692-1700. doi: 10.1016/j.athoracsur.2019.05.079. Epub 2019 Jul 20. PMID 31336066
- See also: Related Info — https://doi.org/10.1016/j.athoracsur.2014.04.110
- See also: Related Info — https://doi.org/10.1016/j.athoracsur.2007.01.048
- See also: Related Info — https://doi.org/10.1186/1749-8090-8-219
- See also: Related Info — https://doi.org/10.1016/j.athoracsur.2019.05.079